CLINICAL TRIAL: NCT02998346
Title: Quantification of Systemic Metabolic Contribution From Continuous Renal Replacement Therapy (CRRT) Utilizing Regional Citrate Anticoagulation
Brief Title: Systemic Metabolic Contribution From Continuous Renal Replacement Therapy (CRRT)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erin Nystrom, Assistant Professor of Pharmacy, Mayo Clinic
Other Study IDs: 13-009155
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Acute Kidney Injury
Keywords: Nutrition; CRRT; CVVH; citrate; anticoagulation; caloric uptake
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to measure the number of calories delivered from fluids used in continuous renal replacement therapy (CRRT). We are doing this research study because the fluids used in this treatment may deliver an important number of calories. In the future this could help better estimate how much nutrition patients in the Critical Care Unit should get every day from other sources like tube feeding or nutrition through a person's veins.

DETAILED DESCRIPTION:
The goal of this study is to quantify the specific metabolic contribution of standard continuous renal replacement protocols (including citrate anticoagulation) in the intensive care unit patient population at Mayo Clinic in Rochester, Minnesota utilizing a prospective, observational study. This data will allow practitioners to better tailor caloric provision with nutrition support programs, minimizing the risk of overfeeding in this complex critical care patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patients in an intensive care unit anticipated to receive greater than or equal to 24 hours of continuous venovenous hemofiltration.
* Receiving regional citrate anticoagulation with ACD-A solution.

Exclusion Criteria:

* Vulnerable adults
* Pregnant
* BMI > 40
* Patient on extracorporeal membrane oxygenation therapy
* Reversal of port connections on the dialysis catheter and dialysis circuit lines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients initiated on continuous venovenous hemofiltration receiving regional citrate anticoagulation with ACD-A solution.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Quantify net glucose uptake from citrate and dextrose-containing fluids from continuous venovenous hemofiltration | Two days
Quantify net citrate uptake from citrate and dextrose-containing fluids from continuous venovenous hemofiltration | Two days

IPD SHARING:
Plan to Share IPD: No